CLINICAL TRIAL: NCT02263404
Title: PINS Stimulator System to Treat Severe Anorexia Nervosa
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINS-004
Record Dates: First submitted 2014-09-27; First posted 2014-10-13 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): DBS Implant and stimulation Intervention: Device: Deep Brain Stimulation
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — DBS Implant Stimulation
  Other Names: Rechargeable Neurostimulator

SUMMARY:
Anorexia Nervosa (AN) has the highest mortality of any psychiatric disorder and a paucity of effective treatments. AN becomes intractable in around 20%, resulting in huge individual and healthcare costs. The study will help patients with severe AN using DBS. Individuals with severe intractable AN will be eligible to take part in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients aged 20-60 years.
2. Diagnosis of anorexia nervosa, restricting or binge-purging subtype, as defi ned in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR).
3. Chronicity or treatment resistance shown by some or all of:

   * A pattern of 3 years' duration of relentless unresponsiveness to repeated voluntary hospital admissions, characterised by failure to complete treatment or immediate weight relapse after treatment.
   * A pattern of increasing medical instability, accompanied by refusal to participate in or a pattern of poor response to intensive expert treatment and increasing medical acuity, lasting at least 2 years and including at least two episodes of involuntary feeding.
   * A pattern of chronic stable anorexia nervosa that has lasted at least 10 years.
   * Able to provide informed consent.
4. Able to comply with all testing, follow-ups, and study appointments and protocols.

Exclusion Criteria:

1. Person with consciousness disorder on opioid abstinence, seriously aggressive, heavily dehydrated and intending to commit suicide.
2. Patients with serious liver and kidney dysfunction, pulmonary decompensation, or complicated with serious damage in other systems.
3. Patients with serious infectious disease.
4. Patients with history of serious neurological or psychiatrical diseases.
5. Person with history of HIV infection or serious malnutrition.
6. Dependent upon and addicted to multiple drugs.
7. Any contraindication to MRI or PET scanning.
8. Body-mass index less than 13.
9. Attended some other trials within one year.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Related Preoccupations and Rituals | Change from baseline in Eating Disorder Related Preoccupations and Rituals scores at 3 months, 6 months and 12 months

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | Change from baseline at 3 months, 6 months and 12 months
Health Survey Short Form (SF-36) | Change from baseline at 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Luming, PhD, Study Chair — Tsinghua University